CLINICAL TRIAL: NCT05462795
Title: Liquid Biopsy to Distinguish Malignant From Benign Pulmonary Nodules and to Monitor Response to Therapy
Brief Title: Liquid Biopsy for Early Non-small Lung Cancer Detection
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2107020697; R43CA257133-01A1 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Non Small-cell Lung Cancer
Keywords: Lung cancer; Biomarker; DNA methylation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Indeterminate pulmonary nodule study cohort: Patients undergoing a biopsy of an indeterminate lung nodule by surgical excision, bronchoscopic biopsy or Interventional Radiology directed biopsy
  Interventions: Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Indeterminate pulmonary nodule
- Known lung cancer for surgical resection study cohort: Patients with known non-small cell lung cancer who will have surgical resection for treatment
  Interventions: Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Known lung cancer for surgical resection
- Healthy volunteer cohort: Healthy volunteers with a) no current diagnosis of cancer; b) no history of cancer over the last 5 years; and c) no existing known benign lung disease that is currently requiring treatment with medication.
  Interventions: Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Healthy volunteer
- Benign lung disease cohort: Patients with the following categories of benign lung disease:
  * COPD/emphysema
  * Granulomatous infection
  * Interstitial lung disease including pulmonary fibrosis and interstitial lung disease.
  Interventions: Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Benign lung disease

INTERVENTIONS:
Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Indeterminate pulmonary nodule — 10 cc of blood is collected at one time point, which is prior to biopsy procedure
  Groups: Indeterminate pulmonary nodule study cohort
Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Known lung cancer for surgical resection — 10 cc of blood is collected at three time points: 1) before surgery; 2) 4-6 weeks post surgery; and 3) 6 months post surgery
  Groups: Known lung cancer for surgical resection study cohort
Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Healthy volunteer — 10 cc of blood is collected at one time point
  Groups: Healthy volunteer cohort
Diagnostic Test: Liquid biopsy for aberrant DNA methylation analysis - Benign lung disease — 30 cc of blood is collected at one time point
  Groups: Benign lung disease cohort

SUMMARY:
This clinical trial will assess the performance of a liquid biopsy assay to identify cancer in indeterminant pulmonary nodules identified by CT screening of high-risk individuals and evaluate the capability of the liquid biopsy assay to monitor response to surgical resection.

DETAILED DESCRIPTION:
This clinical study examines the feasibility of a liquid biopsy methylation assay to detect non-small lung cancer. First, the investigators will apply their liquid biopsy assay to screen for lung cancer in indeterminate pulmonary nodules suspicious for cancer. Second, the investigators will assess the utility of liquid biopsy to assess tumor dynamics after surgical resection with curative intent. Third, the investigators will assess the presence or absence of this methylation assay in healthy normal persons without a history of lung cancer.

ELIGIBILITY:
Indeterminate pulmonary nodule study cohort

* Inclusion criteria: Patients undergoing a biopsy of an indeterminate lung nodule by surgical excision, bronchoscopic biopsy or Interventional Radiology directed biopsy
* Exclusion criteria: No known concurrent cancer

Known lung cancer for surgical resection study cohort

* Inclusion criteria: Patients with known non-small cell lung cancer who will have surgical resection for treatment
* Exclusion criteria: N/A

Healthy volunteer cohort

* Inclusion criteria: Healthy persons
* Exclusion criteria: No known current cancer or history of cancer within 5 years

Benign lung disease cohort

* Inclusion criteria: Patients with the following categories of benign lung disease: COPD/emphysema, Granulomatous infection, Interstitial lung disease including pulmonary fibrosis and interstitial lung disease.
* Exclusion criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and volunteers will be recruited from the BUMC-T Pulmonary and UACC clinics (Indeterminate pulmonary nodule); through study posting on ClinicalTrials.gov and word of mouth (Healthy volunteers); UACC Thoracic Surgery Clinic (Pre-post lung cancer surgery); and Pulmonary Clinic (Benign Lung Disease).
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Indeterminate pulmonary nodule study cohort: Sensitivity and specificity of liquid biopsy test for malignancy | 9 months
  The patients with indeterminate nodules will be used to separately estimate the sensitivity (in those with lung cancer) and specificity (in those without lung cancer). At least 35 patients with lung cancer will provide an estimate of the standard error of the sensitivity < 0.09. Specificity will also be assessed in the normal controls (healthy volunteer cohort) using exact binomial confidence intervals.
Known lung cancer for surgical resection study cohort | 9 months
  To determine the correlation between the longitudinal marker levels and time to progression, to allow adjustment for relevant clinical characteristics.
  Correlations between change in the methylation results and response to therapy using radiographic findings (response, stable disease, progression) at 6 months post-baseline time point will be analyzed using a multinomial regression model.
Healthy volunteers study cohort | 9 months
  Specificity will be assessed in the normal controls (healthy volunteer cohort) using exact binomial confidence intervals.
Benign lung disease cohort | 9 months
  Thirty-five patients with benign lung disease will provide an estimate of the standard error of the specificity <0.09. Assuming a specificity value of 0.91 (32 negative/35 total), the exact 95% confidence interval is (0.77, 0.98). The specificity will be estimated separately, with an exact 95% confidence interval, for each of the benign lung disease subtypes as an exploratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Garland, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No